CLINICAL TRIAL: NCT03511625
Title: The Effects of Acthar on Synovial Inflammation in Rheumatoid Arthritis: A Pilot Study
Brief Title: The Effects of Acthar on Synovial Inflammation in Rheumatoid Arthritis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Attune Health Research, Inc. (Industry)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 32971
Record Dates: First submitted 2018-04-10; First posted 2018-04-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methylprednisolone Acetate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Acthar (Experimental): 80 units of Acthar Injectable Product will be injected subcutaneously daily for three days, followed by twice weekly for four weeks.
  Interventions: Drug: Acthar Injectable Product
- Depo Medrol (Active Comparator): 40 milligrams of Depo Medrol will be injected intramuscularly one time
  Interventions: Drug: Depo medrol

INTERVENTIONS:
Drug: Acthar Injectable Product — Acthar is a non-specific melanocortin receptor agonist
  Other Names: repository corticotropin injection; H.P. Acthar Gel
  Arms: Acthar
Drug: Depo medrol — Depo medrol is an anti-inflammatory glucocorticoid
  Other Names: methylprednisolone acetate injectable suspension
  Arms: Depo Medrol

SUMMARY:
Patients will be assigned to receive either Depo Medrol or Acthar treatment. A synovial biopsy, blood draws, synovial fluid aspiration, and physician assessments will be performed before and after initiating treatment.

DETAILED DESCRIPTION:
Patients will be assigned to receive either Depo Medrol or Acthar treatment. A synovial biopsy, blood draws, synovial fluid aspiration, and physician assessments will be performed before and after initiating treatment. At screening visit, inclusion and exclusion criteria will be assessed. If assessments have not been completed to verify these criteria, they will be performed at this visit. After patients are confirmed to meet criteria, patient disease activity will be assessed and blood draw, synovial aspiration, and biopsy will be performed before first treatment injection. About 5 days after this first treatment injection, these assessment and samples will be performed again. About 5-6 weeks after first treatment injection, a final physician assessment will be performed. Patients will have the option of consenting to allow storage of samples for future research.

ELIGIBILITY:
Inclusion Criteria:

* Anti-Cyclic Citrullinated Peptide positive rheumatoid arthritis
* on a stable regimen of medications
* moderate to severe disease activity as measured by the Clinical Disease activity index (CDAI), or DAS28 (Disease Activity Score) within 30 days of starting the study
* Patients must have at least one joint with the following features within 30 days of starting the study:

  1. Joint must be tender
  2. Joint must be swollen
  3. Joint must have +2 or +3 doppler signal by ultrasound exam
  4. Joint must have +2 or +3 gray scale synovitis by ultrasound exam e. Joint must be amenable to synovial biopsy.

  f. Clinician assessing the joint must conclude, with a reasonable degree of certainty, that the swelling and tenderness observed in the joint is caused by rheumatoid arthritis, and not by another arthritic condition such as osteoarthritis, crystal arthritis, or infection.

Exclusion Criteria:

* Patients on anti-coagulation therapy
* Patients with an active infection
* Patients receiving oral corticosteroids within 5 days of enrollment, or parenteral corticosteroids within 3 weeks of enrollment (unless deemed able to taper off medication under investigator oversight and supervision)
* Patients with any history of joint infection
* Patients with a history of tuberculosis or coccidioidomycosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2018-10-02 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2024-12-03 (Estimated)

PRIMARY OUTCOMES:
Degree of inflammation after short term treatment, as measured by a pathologist during histological assessment | Samples collected about 30 minutes before first treatment injection and about five days after this first injection
  Samples will be sectioned and stained with Haemotoxylin and Eosin and a pathologist blind to treatment will examine the sections under a microscope to determine whether or not inflammation is present compared to how healthy samples would be expected to appear.
Initial degree of inflammation, as measured by a pathologist during histological assessment | Samples collected about five days after first injection of treatment
  Samples will be sectioned and stained with Haemotoxylin and Eosin and a pathologist blind to treatment will examine the sections under a microscope to determine whether or not inflammation is present compared to how healthy samples would be expected to appear.

SECONDARY OUTCOMES:
Initial disease activity as measured by blinded clinician using DAS28 (Disease Activity Score) | Assessments are performed about 1 hour before first treatment injection
  In DAS28, a clinician assesses 28 specified joints for tenderness and swelling. A blood draw is performed at time of assessment to measure Erythrocyte Sedimentation Rate (in mm/h). The patient global health assessment (from 0=best to 100=worst) is also used. A specific algorithm is used to calculate the DAS28 score, using the measurements obtained as variables that plug into the algorithm.
Disease activity after short-term treatment as measured by blinded clinician using DAS28 (Disease Activity Score) | Assessments are performed about 5 days after first treatment injection
  In DAS28, a clinician assesses 28 specified joints for tenderness and swelling. A blood draw is performed at time of assessment to measure Erythrocyte Sedimentation Rate (in mm/h). The patient global health assessment (from 0=best to 100=worst) is also used. A specific algorithm is used to calculate the DAS28 score, using the measurements obtained as variables that plug into the algorithm.
Disease activity after long-term treatment as measured by blinded clinician using DAS28 (Disease Activity Score) | Assessments are performed about 5-6 weeks after first treatment injection.
  In DAS28, a clinician assesses 28 specified joints for tenderness and swelling. A blood draw is performed at time of assessment to measure Erythrocyte Sedimentation Rate (in mm/h). The patient global health assessment (from 0=best to 100=worst) is also used. A specific algorithm is used to calculate the DAS28 score, using the measurements obtained as variables that plug into the algorithm.
Initial number of tender and swollen joints as measured by clinician while palpating 28 specified joints | Assessments are performed about 1 hour before first treatment injection
  A clinician assesses 28 specified joints for tenderness and swelling.
Number of tender and swollen joints after short-term treatment as measured by clinician while palpating 28 specified joints | Assessments are performed about 5 days after first treatment injection
  A clinician assesses 28 specified joints for tenderness and swelling.
Number of tender and swollen joints after long-term treatment as measured by clinician while palpating 28 specified joints | Assessments are performed about 5-6 weeks after first treatment injection.
  A clinician assesses 28 specified joints for tenderness and swelling.
Initial Erythrocyte Sedimentation Rate (ESR) present in blood (in mm/h) | Assessments are performed about 1 hour before first treatment injection
  The Westergren method requires collecting 2 ml of venous blood into a tube containing 0 .5 ml of sodium citrate. It should be stored no longer than 2 hours at room temperature or 6 hours at 4 °C. The blood is drawn into a Westergren-Katz tube to the 200 mm mark. The tube is placed in a rack in a strictly vertical position for 1 hour at room temperature, at which time the distance from the lowest point of the surface meniscus to the upper limit of the red cell sediment is measured. The distance of fall of erythrocytes, expressed as millimeters in 1 hour, is the Erythrocyte Sedimentation Rate.
Erythrocyte Sedimentation Rate (ESR) present in blood (in mm/h) after short-term treatment | Assessments are performed about 5 days after first treatment injection
  The Westergren method requires collecting 2 ml of venous blood into a tube containing 0 .5 ml of sodium citrate. It should be stored no longer than 2 hours at room temperature or 6 hours at 4 °C. The blood is drawn into a Westergren-Katz tube to the 200 mm mark. The tube is placed in a rack in a strictly vertical position for 1 hour at room temperature, at which time the distance from the lowest point of the surface meniscus to the upper limit of the red cell sediment is measured. The distance of fall of erythrocytes, expressed as millimeters in 1 hour, is the Erythrocyte Sedimentation Rate.
Erythrocyte Sedimentation Rate (ESR) present in blood (in mm/h) after long-term treatment | Assessments are performed about 5-6 weeks after first treatment injection.
  The Westergren method requires collecting 2 ml of venous blood into a tube containing 0 .5 ml of sodium citrate. It should be stored no longer than 2 hours at room temperature or 6 hours at 4 °C. The blood is drawn into a Westergren-Katz tube to the 200 mm mark. The tube is placed in a rack in a strictly vertical position for 1 hour at room temperature, at which time the distance from the lowest point of the surface meniscus to the upper limit of the red cell sediment is measured. The distance of fall of erythrocytes, expressed as millimeters in 1 hour, is the Erythrocyte Sedimentation Rate.
Initial patient global health assessment measured by the patient (from 0=best to 100=worst) | Assessments are performed about 1 hour before first treatment injection
  A patient is asked to rate their general global health on a scale from 0 to 100
Patient global health assessment measured by the patient (from 0=best to 100=worst) after short-term treatment | Assessments are performed about 5 days after first treatment injection
  A patient is asked to rate their general global health on a scale from 0 to 100
Patient global health assessment measured by the patient (from 0=best to 100=worst) after long-term treatment | Assessments are performed about 5-6 weeks after first treatment injection.
  A patient is asked to rate their general global health on a scale from 0 to 100

CONTACTS AND LOCATIONS:
Overall Officials: Swamy R Venuturupalli, MD, FACR, Principal Investigator — CEO
Locations (1):
- Attune Health, Beverly Hills, California, United States